CLINICAL TRIAL: NCT05122663
Title: A Pilot Feasibility Trial of Emergency Department Vestibular Rehabilitation Therapy for Dizziness and Vertigo
Brief Title: Emergency Department Vestibular Rehabilitation Therapy for Dizziness and Vertigo
Acronym: ED-VeRT
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Howard Kim, Assistant Professor, Northwestern University
Other Study IDs: STU00215925
Record Dates: First submitted 2021-11-12; First posted 2021-11-17 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Dizziness; Vertigo
MeSH Terms: conditions — Dizziness; Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ED Physical Therapy: Patients in the ED physical therapy group will have been evaluated by an emergency department physical therapist for dizziness/vertigo during their index ED visit.
  Interventions: Behavioral: Vestibular Rehabilitation
- Usual Care: Patients in the usual care group will NOT have received an evaluation by an ED physical therapist for dizziness/vertigo symptoms during their index ED visit.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Vestibular Rehabilitation — Vestibular Rehabilitation refers to the specific interventions that physical therapists provide to patients with dizziness and vertigo symptoms. These interventions can involve repositioning maneuvers, habituation exercises, gaze stabilization, and/or balance training exercises, depending on the specific etiology of dizziness and vertigo per an established clinical protocol utilizing a patient's history and exam findings. Physical therapists instruct patients in how to perform these exercises at home and provide instructions and referral for patients to follow-up with an outpatient physical therapist for further care.
  Groups: ED Physical Therapy
Other: Usual Care — Usual Care refers to any combination of diagnostic testing, medications, and patient education or counseling provided by a patient's treating ED physician.
  Groups: Usual Care

SUMMARY:
ED-VeRT will enroll up to 125 adult emergency department (ED) patients presenting with a chief complaint of dizziness or vertigo to collect longitudinal outcomes over 3 months of follow-up. This will include 50 patients who were evaluated by an ED physical therapist (ie, vestibular rehabilitation) during their ED visit and 50 patients who received usual care. The aims of this trial are to: (1) obtain initial estimates of participant recruitment and retention, intra-cluster correlation, and between-group outcome differences that will inform sample size calculation for a future randomized clinical trial, and (2) assess feasibility and fidelity of a clinical classification protocol for undifferentiated dizziness among patients receiving ED vestibular rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint relating to dizziness or vertigo
* Ability to complete follow-up data collection electronically or by telephone
* English-speaking

Exclusion Criteria:

* Severe neurologic deficit concerning for ischemic or hemorrhagic stroke
* Known pregnancy, under police custody, unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ED patients presenting with a chief complaint relating to dizziness or vertigo.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory (DHI) | Three months after the index ED visit.
  The DHI contains 25 items quantifying self-perceived handicapping effects of dizziness symptoms.

SECONDARY OUTCOMES:
Vestibular Activities Avoidance Instrument (VAAI-9) | Three months after the index ED visit.
  The VAAI-9 identifies fear avoidance beliefs in persons with dizziness. The VAAI-9 is the 9-item short form version of the VAAI.
ED Diagnostic Imaging Utilization | Index ED visit (one day)
  The proportion of ED visits in which any diagnostic imaging of the brain was performed, including computed tomography and magnetic resonance imaging.
ED Length of Stay | Index ED visit (up to one week)
  Total length of stay, inclusive of hospitalizations and observation stays.
Patient-Reported Medication Use in Last 24 Hours | Three months after the index ED visit.
  Patient-reported medication use for dizziness will be collected using a standardized instrument assess whether participants have taken any dizziness medication in the last 24 hours (binary yes/no). The 24-hour timeframe was selected to maximize accuracy in patient recall. In brief, dizziness medications are listed by brand and generic names; a "yes" response to any medication triggers an additional query asking the participant to specify the medication dose (e.g., meclizine 25mg) and quantity (e.g., one pill).

OTHER OUTCOMES:
Global Rating of Change (GROC) | Three months after the index ED visit.
  The GROC is a single-item survey used to evaluate overall recovery from the time that symptoms began until now. Responses are provided on a 15-point Likert scale ranging from "a very great deal worse" to "a very great deal better."
Numeric Rating Scale (NRS) | Three months after the index ED visit.
  The NRS measures intensity of dizziness symptoms from 0 to 10. Participants will report average dizziness intensity over the last 24 hours.
Advanced Healthcare Utilization | Three months after the index ED visit.
  Proportion of participants who utilized any advanced healthcare resources for dizziness after their index ED visit, defined as advanced imaging (e.g., computed tomography, magnetic resonance imaging) or procedures/surgery.
Benzodiazepine Prescription Filling | Three months after the index ED visit
  Benzodiazepine prescription filling data will be queried in the state prescription monitoring database.
Follow-up with Outpatient Physical Therapy | Three months after the index ED visit
  Proportion of participants who reports outpatient physical therapy follow-up for vestibular rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HS, Schauer JM, Kan AK, Alinger JB, Strickland KJ, Garreau A, McCarthy DM, Taylor ZB, Fishman IL, Muschong KM, Roth HR. Emergency Department Vestibular Rehabilitation Therapy for Dizziness and Vertigo: A Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2459567. doi: 10.1001/jamanetworkopen.2024.59567. PMID 39951266

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT05122663/SAP_000.pdf